CLINICAL TRIAL: NCT04713189
Title: A Phase I/IIa, Pharmacokinetic, Dose-response and Safety Study of Inhaled Fentanyl Aerosol (25µg/Dose) in Chinese Patients With Breakthrough Cancer Pain
Brief Title: Effectiveness and Tolerance of Inhaled Fentanyl Aerosol (25µg/Dose) in Chinese Patients With Breakthrough Cancer Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZK05
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Breakthrough Cancer Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled fentanyl aerosol (Experimental): Participants in the stage I were randomized to 6 BTP episodes, in which 4 BTP episodes were treated with inhale fentanyl aerosol (with a starting dose of 25 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×25 µg) and 2 BTP episodes with placebo(0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence.
  Interventions: Drug: Inhaled fentanyl aerosol
- Placebo (Experimental): Participants in the stage I were randomized to 6 BTP episodes, in which 2 BTP episodes were treated with placebo (0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled fentanyl aerosol — Participants in the stage I were randomized to 6 BTP episodes, in which 4 BTP episodes were treated with inhale fentanyl aerosol (with a starting dose of 25 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×25 µg) and 2 BTP episodes with placebo(0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence.
  Arms: Inhaled fentanyl aerosol
Drug: Placebo — Participants in the stage Ⅰ were randomized to 6 BTP episodes, in which 2 BTP episodes were treated with placebo (0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence. I
  Arms: Placebo

SUMMARY:
Breakthrough cancer pain (BTcP) is a common problem in patients with cancer. This is a phase I/IIa, pharmacokinetic, dose-response and safety study of inhaled fentanyl aerosol (25µg/dose) in Chinese patients with breakthrough cancer pain. The study will include two stages.

DETAILED DESCRIPTION:
Stage I: dose-response relationship and safety assessment of inhaled fentanyl aerosol in patients with breakthrough cancer pain. placebo-controlled, cross-over, double-blind randomized design is applied in this stage.

Patients meeting the inclusion/exclusion criteria will be treated with inhaled fentanyl aerosol (4 of 6 episodes BTcp) or placebo (2of 6 episodes BTcp).Subjects will inhale fentanyl aerosol or placebo for each episode of BTcp with a starting dose of 25 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×25 µg.

Stage II: The dosage regimen (number of puffs) will be depended on the data from Stage I. Subjects will inhale fentanyl aerosol not in the episode of breakthrough cancer pain with a starting dose of 25 µg every 4 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 75years, inclusive.
2. Subjects must be diagnosed with cancer.
3. Subjects must be opioid-tolerant : taking oral morphine more than 60mg and less than 1000mg,or taking other equivalent potency opioids of analgesic doses in one weeks or longer.
4. Subjects must experience persistent pain associated with cancer, and the pain score assessed by NRS should be <4 within 24hour before screening.
5. The breakthrough cancer pain score should be ≥4 assessed by NRS.
6. In the past 7 days, the subject must experience an average of 1 to 4 episodes of breakthrough cancer pain per day, and use 5 mg immediate release morphine at least or equivalent short-acting opioids (e.g., oxycodone, hydrocodone ketones or codeine) to control this pain.
7. ECOG status of 0 to 2.
8. Life expectancy should be longer than 3 months.
9. Subjects must consent to take adequate contraception within the study and 1 months after the study. Women of childbearing potential must show negative in the pregnancy test before dosing.
10. The subject must be able to understand the requirements of the study and provide a written informed consent.

Exclusion Criteria:

1. Allergies, or a history of drug allergies to fentanyl.
2. On intrathecal or epidural opioids.
3. HGB < 80 g/L, NEUT ≤1.5 × l09/L, PLT ≤50 × l09/L；ALT and AST higher than 3 times of ULN;total bilirubin and Cr higher than 1.5 times of ULN;PaO2 <95%;FEV1/FVC<70% and FEV1 accounted for less than 80% of the predicted value.
4. Any uncontrolled disease (e.g., severe mental, neurological, infectious, cardiovascular, respiratory and other systemic diseases).
5. Hepatitis B surface antigen and hepatitis C surface antibody positive. Human T Lymphotropic Virus Type I Positive. HIV positive.
6. Gastrointestinal bleeding or diarrhea presently.
7. Requirement of continuous paracentesis.
8. Tumor infiltration to central nervous system.
9. Subjects are not able to slef evaluate pain intensity using NRS
10. Receive surgery in past 3 weeks.
11. Treatment with any form of radiotherapy winth 1week prior to study entry that could alter pain or response to pain medication.
12. Taking monoamine oxidase inhibitors(MAOIs), CYP3A4 inhibitors or inducers within 14 days of the screening
13. Participated in other clinical trials in past 1months.
14. Pregnancy and breast-feeding women, women of childbearing age ready to conceive, and pregnancy test positive.
15. Other conditions that may affect the informed consent, compliance with the protocol, study results and safety of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-12-21 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
SPID30 | During the stage I, at each episode of breakthrough pain, 30 minutes after first dose of study drug.
  Weighted sum of pain intensity difference at post dose 30 minutes.Pain intensity at each breakthrough pain (BTP) episode at 0 ,4,8,12,16,20 and 30 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID30 is calculated as the difference in pain intensity from time 0 to 30 minutes. A positive value is a decrease (improvement) of the pain.SPID30=PID4*4+PID8*4+PID12*4+PID16*4+PID20*4+PID30*10

SECONDARY OUTCOMES:
Pain intensity at 0, 4,8,12,16,20,30 and 60 minutes post-dose | During the stage I, at each episode of breakthrough pain, 60 minutes after first dose of study drug.
  Pain intensity at each breakthrough pain (BTP) episode at 0 ,4,8,12,16,20, 30 and 60 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain".A positive value is a decrease (improvement) of the pain.
SPID60 | During the stage I, at each episode of breakthrough pain, 60 minutes after first dose of study drug.
  Weighted sum of pain intensity difference at post dose 60 minutes.Pain intensity at each breakthrough pain (BTP) episode at 0 ,4,8,12,16,20, 30 and 60 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID60 is calculated as the difference in pain intensity from time 0 to 60 minutes. A positive value is a decrease (improvement) of the pain.SPID60=PID4*4+PID8*4+PID12*4+PID16*4+PID20*4+PID30*10+PID30*30
Percentage of episodes with NRS≤3 | Through study completion, an average of 4 days
  Overall responder rate is defined as the proportion of breakthrough pain (BTP) episodes with a positive response to treatment. The following definitions of a positive response were analyzed: greater than or equal to 3 point reduction in PI from time 0. Pain intensity was assessed using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain".
Percentage of episodes with at least 33% and 50%decrease in pain | Through study completion, an average of 4 days
  Overall responder rate is defined as the proportion of breakthrough pain (BTP) episodes with a positive response to treatment. The following definitions of a positive response were analyzed: Greater than 33% reduction in PI from time 0;Greater than 50% reduction in PI from time 0. Pain intensity was assessed using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain".
Rescue medication usage | Through study completion, an average of 4 days
  Only Morphine for injection to be used as rescue medication

OTHER OUTCOMES:
device performance | through study completion, an average of 4 days
  Success rate of drug stimulation (successful drug inhalation). Normal rate of electronic lock function.

REFERENCES:
- [Derived] Lin R, Song B, Li N, Rong B, Bai J, Liu Y, Wang W, Liu A, Luo S, Liu B, Cheng P, Wu Y, Li Y, Yu X, Liu X, Dai X, Li X, Liu D, Wang J, Huang Y. Efficacy and safety of fentanyl inhalant for the treatment of breakthrough cancer pain: a multicenter, randomized, double-blind, placebo-controlled trial. BMC Palliat Care. 2024 Sep 7;23(1):222. doi: 10.1186/s12904-024-01554-9. PMID 39244530